CLINICAL TRIAL: NCT06017661
Title: Investigation of a Polyphenol-rich Preparation as Support for Oncology Patients Undergoing Gastrointestinal Tumor Resection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: AronPharma Sp. z o. o. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 09-AP-ONCON
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-08

CONDITIONS: Immunomodulation
Keywords: chokeberry; Nutridrink; immunomodulation; tumor resection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nutridrink Skin Repair with a mixture of plant extracts rich in polyphenolic compounds (Experimental): Group of 15 patients undergoing surgical resection of tumour
  Interventions: Dietary Supplement: Nutridrink Skin Repair with a mixture of plant extracts rich in polyphenolic compounds
- Nutridrink Skin Repair (Active Comparator): Group of 15 patients undergoing surgical resection of tumour
  Interventions: Dietary Supplement: Nutridrink Skin Repair

INTERVENTIONS:
Dietary Supplement: Nutridrink Skin Repair with a mixture of plant extracts rich in polyphenolic compounds — 2 times a day
  Arms: Nutridrink Skin Repair with a mixture of plant extracts rich in polyphenolic compounds
Dietary Supplement: Nutridrink Skin Repair — 2 times a day
  Arms: Nutridrink Skin Repair

SUMMARY:
The aim of the study is to demonstrate, under clinical conditions, the effectiveness of the standard product 'Nutridrink' enriched with a mixture of plant extracts rich in polyphenolic compounds in the aspect of supporting the recovery of oncology patients undergoing surgical resection of tumours.

DETAILED DESCRIPTION:
Oncology patients undergoing the procedure are exposed to various postoperative complications. Nutridrink with a mixture of extracts with anti-inflammatory and antioxidative properties aims to provide the patient with essential nutrients and bioactive substances that can reduce the inflammatory state, protect cells from oxidative damage, and decrease the risk of complications while supporting tissue healing processes after the surgical procedure. The study group are oncology patients undergoing surgical resection of gastrointestinal tumour. During the study, the effects of the mixture on levels of oxidative stress and inflammation markers will be assessed, as well as the subjective evaluation of patients' quality of life and well-being after surgical surgical tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* Women and men, 18-80 years old
* Patients diagnosed with resectable gastrointestinal tract cancer undergo the resection procedure no later than one month after being enrolled in the study
* Signed informed consent

Exclusion Criteria:

* Intake of supplements containing plant extracts, polyphenols or anthocyanins
* Participation in another clinical trial
* Inability to consume the investigational product in liquid form as medication/placebo
* Women who are pregnant, planning to become pregnant during the study or breastfeeding
* Autoimmune disease, severe liver dysfunction, inflammatory bowel disease, tuberculosis, multiple sclerosis, AIDS, rheumatoid arthritis, organ transplantation
* Hypersensitivity/allergy to any of the ingredient

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-12-15 (Estimated); Study Completion 2023-12-15 (Estimated)

PRIMARY OUTCOMES:
SOD level | Baseline, 3 weeks, 6 weeks
  Comparison of SOD level
GSH level | Baseline, 3 weeks, 6 weeks
  Comparison of GSH level
IL-6 level | Baseline, 3 weeks, 6 weeks
  Comparison of IL-6 level
IL-8 level | Baseline, 3 weeks, 6 weeks
  Comparison of IL-8 level

SECONDARY OUTCOMES:
Patients' quality of life | Baseline, 3 weeks, 6 weeks
  Subjective assessment of patients' quality of life after surgical resection of the tumor (questionnaire). Higher scores mean a better outcome.

CONTACTS AND LOCATIONS:
Locations (1):
- Uniwersyteckie Centrum Kliniczne, Klinika Chirurgii Onkologicznej, Transplantacyjnej i Ogólne, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No